CLINICAL TRIAL: NCT01014780
Title: Tear Film Thickness Measured Using a Novel Technique
Status: Completed | Type: Observational
Sponsor: Southern California College of Optometry at Marshall B. Ketchum University (Other)
Responsible Party: Jerry R. Paugh, Southern California College of Optometry
Other Study IDs: 09-10
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Last update posted 2010-10-11 (Estimated); Status verified 2010-09

CONDITIONS: Dry Eye
Keywords: dry eye; tear film; thickness; artificial tears
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal (non-dry) dry eye subjects: These are healthy individuals, age 18 and above, who do not exhibit dry eyes by signs and symptoms
- Dry eye subjects: These are subjects, age 18 years and above, who do exhibit signs and symptoms of dry eye.

SUMMARY:
The aim of this investigation is to determine the thickness of the human preocular tear film using a new method based on laser speckle. This will be a preliminary study to generate "normative" tear film thickness data in normal (i.e., non dry eye) and dry eye subjects in a clinic-based population. In addition, we will examine the short term (i.e., one week) repeatability of the method in a single setting.

The patients classified as having dry eye will also have their tear film thickness measured after instillation of an artificial tear. This will potentially reveal valuable data in retention of effect measured non-invasively as in prior studies that employed a fluorescein tracer.

DETAILED DESCRIPTION:
We will generate "normative" tear thickness data in normal (i.e., not dry) and dry eyes in human subjects. We will examine short-term repeatability of the method, and we will examine the influence on tear thickness of a viscous eyedrop instilled into the eye.

ELIGIBILITY:
Inclusion Criteria:

There are no requirements as to subject race, gender or occupation. If the subjects have any questions or concerns regarding any of the inclusion or exclusion criteria, they will be encouraged to ask either investigator (Dr. Paugh or Dr. Kwan) for clarification. All subjects must meet the following criteria:

1. The informed consent document must be read, signed and dated by the subject before conducting any procedures. Additionally, the informed consent document must be signed and dated by the individual obtaining consent of the subject. HIPAA authorization must also be signed and dated by the subject.
2. Adult subjects, 18 years of age and older. Criteria for the mild to severe dry eye group must include two of the three following characteristics as demonstrated at the Eligibility visit:

   1. Composite symptom score of ≥ 7 on the Schein questionnaire:
   2. Sodium fluorescein (NaFl) tear break-up time ≤ 7 seconds in either (worse) eye
   3. Cumulative sodium fluorescein (NaFl) corneal staining ≥ 4 in either (worse) eye on a 0-20 point scale (corresponds to ≥ 3.0 on a 0-15 scale).
3. Able and willing to follow study instructions.
4. Willing to return for the repeatability visit within 7 plus or minus 2 days of the initial visit, and within the same one-half day (i.e., either in the morning or afternoon, similar to the first tear thickness visit).
5. Subjects must have best corrected visual acuity of 20/25 or better in each eye as assessed using a standard Snellen acuity chart.
6. Subjects wearing soft contacts lenses must be willing to discontinue wear for two days before each study visit.
7. Subjects using any topical drops such as artificial tears must be willing to discontinue use of such drops for two days prior to all visits, including the baseline visit.

Exclusion Criteria:

Subjects demonstrating any medical condition that may affect the results of this study SHOULD NOT be enrolled. The following are specific conditions that exclude subjects from enrollment in this study:

1. History or evidence of ocular or intraocular surgery in either eye within the past six months. LASIK and other kerato-refractive procedure patients can qualify if the most recent surgery or enhancement was 12 or more months prior.
2. History or evidence of serious ocular trauma in either eye within the past six months.
3. History of hypersensitivity to sodium fluorescein.
4. History or evidence of epithelial herpes simplex keratitis (dendritic keratitis); vaccinia, active or recent varicella, viral disease of the cornea and/or conjunctiva; chronic bacterial disease of the cornea and/or conjunctiva; mycobacterial infection of the eye; and/or fungal disease of the eye.
5. Patients requiring use of topical ocular medications such as glaucoma or allergy medications during the study period.
6. Individuals using systemic steroids, immunosuppressive agents and/or anti-cholinergics (e.g. cold and allergy medications, tricyclic antidepressants) for treatment of autoimmune connective tissue disease may not be enrolled in the study if they have not been on a stable dosing regimen for a minimum of 30 days prior to the first visit. In addition, the dosing regimen must remain stable throughout the study period, expected to be approximately one week.
7. Individuals with diabetes.
8. Ocular conditions such as conjunctival infections, or iritis.
9. Individuals wearing rigid gas permeable contact lenses or using punctal plugs.
10. Participation in an investigational drug or device study within 30 days of entering this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will inculde up to 20 normals (i.e., non-dry eye) individuals, over the age of 18 years, adn 20 dry eye individuals.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-04 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Tear film thickness in normal eyes | 1-3 months

SECONDARY OUTCOMES:
Tear thickness change following viscous drop instillation | 1-3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Paugh, OD. PhD, Study Director — Southern California College of Optometry at Marshall B. Ketchum University
Locations (1):
- Southern California College of Optometry, Fullerton, California, United States